CLINICAL TRIAL: NCT04399434
Title: Study on the Relationship of Gut Microbiota and Changes of SCFAs With Glucolipid Metabolism in Pregnant Women With Abnormal Fetal Size and Their Newborns
Brief Title: Gut Microbiota, SCFAs and Glucolipid Metabolism in Pregnant Women With Abnormal Fetal Size and Their Newborns
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2020-07-209
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Fetal Growth Restriction; Gut Microbiota; Fetal Macrosomia; Glucolipid Metabolism
MeSH Terms: conditions — Fetal Growth Retardation; Fetal Macrosomia | interventions — Insulin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- normal pregnancy: pregnancy with a normal fetal size
  Interventions: Other: test gut microbiota, SCFAs and glucolipid metabolism and insulin sensitivity
- fetal growth restriction: fetal birth weight is below two standard deviations of the average weight for the same gestational age, or below the 10th percentile of normal weight for the same age
  Interventions: Other: test gut microbiota, SCFAs and glucolipid metabolism and insulin sensitivity
- fetal macrosomia: fetal birth weight ≥ 4000g
  Interventions: Other: test gut microbiota, SCFAs and glucolipid metabolism and insulin sensitivity

INTERVENTIONS:
Other: test gut microbiota, SCFAs and glucolipid metabolism and insulin sensitivity — test gut microbiota and SCFAs in mothers and their newborns and glucolipid metabolism and insulin sensitivity in mothers

SUMMARY:
Abnormal fetal size includes fetal growth restriction and fetal macrosomia. Onset is closely related to maternal nutrition metabolism. The specific correlation and mechanism is unclear, and there are no effective measures for early diagnosis and treatment. Previous study found that maternal gut microbiota participates in the material metabolism throughout the pregnancy. Insulin sensitivity in pregnant women, and intrauterine environment under abnormal blood glucose and lipid metabolism are important for the gut microbiota of newborns and even they grow up. However, changes in gut microbiota are the cause of the disease or the outcome is not yet clear. Short chain fatty acids (SCFAs) are produced from soluble dietary fibers in the diet by colon bacteriolysis. Studies have found that gut microbiota can regulate insulin sensitivity and glucose and lipid metabolism disorders through SCFAs. Therefore, this research group uses the gut microbiota as a new idea to studythe relationship of gut microbiota characteristics and level's change of SCFAs with glucolipid metabolism and insulin sensitivity in pregnant women with abnormal fetal size and their newborns through 16S-rRNA high-throughput sequencing, pyrosequencing, and gas chromatography-mass spectrometry, so we can reveal the role of gut microbiota in the pathogenesis of abnormal fetal size and explore targeted rational dietary adjustment and SCFAs reconstruction of gut microbiota to improve maternal and neonatal pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Term pregnancy with the gestational age of 37-40 weeks

Exclusion Criteria:

* Maternal systemic diseases (hypertension disorders, immunological diseases) or pregnant complications (polyhydramnios, oligohydramnios, diabetes mellitus, intrahepatic cholestasis of pregnancy)
* Delivery before 37 weeks or after 40 weeks
* Neonates had major congenital malformations (congenital anal atresia, congenital biliary atresia, congenital heart disease)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligible participants is female.
Study Population: The participants include mother-infant pairs meeting the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiota and SCFAs in mothers and their newborns | Stool samples from pregnant women with 37-40 gestational week and newborns within 3 days after birth
  Collect the DNA of fecal flora to test the diversity and abundance of gut microbiota as well as short chain fatty acids in Stool samples
glucolipid metabolism and insulin sensitivity in pregnant women | Blood samples from pregnant women with 37-40 gestational week
  glucolipid metabolism and insulin sensitivity in pregnant women with normal and abnormal fetal size

CONTACTS AND LOCATIONS:
Overall Officials: Ying Hua, Study Director — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- department of obstetrics of Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China